CLINICAL TRIAL: NCT04949282
Title: SEPTRALU, Spanish Series of Patients Treated With the Radionuclide Lutetium177
Brief Title: Spanish Series of Patients Treated With the Radionuclide Lutetium177
Acronym: SEPTRALU
Status: Recruiting | Type: Observational
Sponsor: Sociedad Española de Medicina Nuclear e Imagen Molecular (Other)
Responsible Party: Sponsor
Other Study IDs: SEM-LUT-2020-01
Record Dates: First submitted 2021-06-14; First posted 2021-07-02 (Actual); Last update posted 2022-12-23 (Actual); Status verified 2022-12

CONDITIONS: Neuroendocrine Tumors; Intestinal Neoplasms; Pancreatic Neoplasms; Stomach Neoplasms; Neuroectodermal Tumors; Neoplasms, Germ Cell and Embryonal; Neoplasms by Histologic Type; Neoplasms; Neoplasms, Nerve Tissue; Gastrointestinal Neoplasms; Digestive System Neoplasms; Neoplasms by Site; Endocrine Gland Neoplasms; Digestive System Diseases; Gastrointestinal Disease; Intestinal Diseases; Pancreatic Disease; Endocrine System Diseases
Keywords: GEP-NET; Gastro-Entero-Pancreatic Neuroendocrine Tumour; Luthatera; Somatostatin receptor positive tumour
MeSH Terms: conditions — Neuroendocrine Tumors; Intestinal Neoplasms; Pancreatic Neoplasms; Stomach Neoplasms; Neuroectodermal Tumors; Neoplasms, Germ Cell and Embryonal; Neoplasms by Histologic Type; Neoplasms; Neoplasms, Nerve Tissue; Gastrointestinal Neoplasms; Digestive System Neoplasms; Neoplasms by Site; Endocrine Gland Neoplasms; Digestive System Diseases; Gastrointestinal Diseases; Intestinal Diseases; Pancreatic Diseases; Endocrine System Diseases; Gastro-enteropancreatic neuroendocrine tumor | interventions — Lutetium; Lutetium-177; copper dotatate CU-64; lutetium Lu 177 dotatate

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Lutathera
  Interventions: Drug: Lutetium [177Lu] oxodotreotide/dotatate; Device: Lutetium [177Lu] oxodotreotide/dotatate

INTERVENTIONS:
Drug: Lutetium [177Lu] oxodotreotide/dotatate — Radiopharmaceutical solution for infusion (7.4 GBq of Lutathera per 30 ml vial)
  Other Names: Lutathera
Device: Lutetium [177Lu] oxodotreotide/dotatate — Radiopharmaceutical solution for infusion (7.4 GBq of Lutathera per 30 ml vial)
  Other Names: Lutathera

SUMMARY:
This study aims to pool the clinical experience of Spanish centers treating patients with 177Lu-DOTATATE to evaluate the efficacy, tolerance, and safety of the drug in routine clinical practice and to learn about the profiles of patients and tumors treated and the results in each type of patient and tumor.

DETAILED DESCRIPTION:
Patient data will be collected from medical records after obtaining consent and retrospectively.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent must be obtained prior to any data collection.
* Patients must be diagnosed with unresectable or metastatic, progressive, somatostatin receptor positive tumour
* Aged ≥18 years.

Exclusion Criteria:

* None

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study plans to enroll patients with unresectable or metastatic, progressive, somatostatin receptor positive tumors.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2021-05-10 (Actual); Primary Completion 2034-12-31 (Estimated); Study Completion 2035-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | Up to 12 months
  Defined as the time, in months, from Lutathera® treatment initiation to the date of first objective tumour progression, determined according to Response Evaluation Criteria in Solid Tumours (RECIST) Criteria, Version 1.1, or death due to any cause, whichever comes first.
Overall survival (OS) | Up to 12 months
  Defined as the time, in months, from Lutathera® treatment initiation to the date of death due to any cause.
Overall response rate (ORR) | Up to 12 months
  Is determined by imaging technique according to RECIST criteria v1.1 and is defined as the proportion of treated patients who achieve a best overall response of partial response (PR) or complete response (CR) according to RECIST 1.1

SECONDARY OUTCOMES:
Characteristics of the population . | Up to 12 months
  Description of the main characteristics of the population studied, treatments received (before and after lutetium) and evolution.
Adverse Events (AEs) | Up to 12 months
  Toxicity will be collected according to grades (NCT-CTCAE) and consequences.
Prognostic factors | Up to 12 months
  Correlation of possible prognostic factors with clinical effectiveness outcomes.
Areas for improvement care | Up to 12 months
  Identification of areas for improvement in the management and selection of patients for treatment with lutathera
Health-related Quality of Life (HRQoL) | Up to 12 months
  Assess the impact of treatment on health-related Quality of Life (HRQoL) by EORTC QLQ-G.I.NET-21 questionnaire.The minimum value ( 1%) and the maximum value (100%), and higher scores mean a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Mercedes Dr Mitjavila Casanovas, MD-PhD, Principal Investigator — Sociedad Española de Medicina Nuclear e Imagen Molecular (SEMNIM)
Locations (20):
- Spain (20):
  - Hospital Clínico Universitario de Santiago, Santiago de Compostela, A Coruña
  - Hospital Universitario Virgen de las Nieves, Granada, Andalusia
  - Hospital Unviersitari Son Espases, Palma de Mallorca, Balearic Islands
  - Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario de Getafe, Getafe, Madrid
  - Hospital Univeritario Puerta de Hierro, Majadahonda, Madrid
  - Hospital Clínico Universitario Virgen de la Arrixaca, El Palmar, Murcia
  - Clínica Universidad de Navarra, Pamplona, Navarre
  - Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario de Burgos, Burgos
  - Hospital General Universitario de Ciudad Real, Ciudad Real
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario HM Sanchinarro, Madrid
  - Hospital Universitario de Navarra, Pamplona
  - Hospital Universitario Doctor Peset, Valencia
  - Hospital Universitario La Fe, Valencia

REFERENCES:
- [Derived] Mitjavila M, Jimenez-Fonseca P, Bello P, Pubul V, Percovich JC, Garcia-Burillo A, Hernando J, Arbizu J, Rodeno E, Estorch M, Llana B, Castellon M, Garcia-Canamaque L, Gajate P, Riesco MC, Miguel MB, Balaguer-Munoz D, Custodio A, Cano JM, Repetto A, Garcia-Alonso P, Muros MA, Vercher-Conejero JL, Carmona-Bayonas A. Efficacy of [177Lu]Lu-DOTATATE in metastatic neuroendocrine neoplasms of different locations: data from the SEPTRALU study. Eur J Nucl Med Mol Imaging. 2023 Jul;50(8):2486-2500. doi: 10.1007/s00259-023-06166-8. Epub 2023 Mar 6. PMID 36877234